CLINICAL TRIAL: NCT06433570
Title: Detection of Krupple Like Factor -1(KLF1/ EKLF) DNA Mutations in Beta Thalassemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elnasser Mahmoud, Assiut, Assiut University
Other Study IDs: EKLFmutation in β thalassemia
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: EKLF Mutations in Beta Thalassemia Patients
MeSH Terms: interventions — Multiplex Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 patients with beta thalassemia intermedia
  Interventions: Genetic: multiplex PCR
- 50 patients with beta thalassemia major
  Interventions: Genetic: multiplex PCR

INTERVENTIONS:
Genetic: multiplex PCR — Detection of Krupple Like Factor -1(KLF1/ EKLF) DNA Mutations in Beta Thalassemia Patients using multiplex PCR

SUMMARY:
* Detection of KLF1 gene mutations in patients with beta thalassemia considering the alpha and beta molecular status of these patients.
* Study the relation between genotypic mutational status of KLF1 mutation with the level of Hb F and Hb A2 in the patients of beta thalassemia.

DETAILED DESCRIPTION:
Thalassemias are inherited abnormalities in globin chain synthesis of hemoglobin and one of the most common single gene disorders in the world.

β-Thalassemia is caused by reduced (β+) or absent (β0) synthesis of the β-globin chains of haemoglobin. Three clinical and hematological conditions of increasing severity are recognized: the β-thalassemia trait, thalassemia intermedia and thalassemia major.

The Erythroid Kruppel-like factor (EKLF or KLF1) is a master regulator of terminal erythroid differentiation, controlling expression of many key pathways and structures including cell division, the cell membrane and cytoskeleton, heme and globin synthesis.

The KLF1 works as a key regulator of γ-globin to β-globin switch by up-regulation of PUM1 that binds to fetal γ globin mRNA impairing its stability and translation and by Bcl11a expression that represses γ-globin expression.

Previous studies reported that KLF1 mutations have been identified in a variety of erythroid conditions like hereditary persistence of fetal hemoglobin, Congenital dyserythropoietic anemia and borderline HbA2.

An Indian study on KLF1 gene variations found a marginal significance in the thalassemia intermedia group (14%) as against the thalassemia major group (2.0%).

Also, a case report on a Chinese family with twin brothers, both of whom had the same genotype of β0/β0, reported that KLF1 mutations have a role in modulating the phenotypic severity of β-thalassemia.

In our study, where there is high incidence of beta thalassemia in Egypt, we try to detect KLF1 mutations and its relation to clinical phenotype of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with β-thalassemia (intermedia and major) of both genders at any age

Exclusion Criteria:

* Patients with any other type of haemolytic anaemias.
* Patients on Hydroxyurea therapy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: cross sectional study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Detection of KLF1 gene mutations in patients with beta thalassemia considering the beta molecular status of these patients | Baseline
  Study the relation between genotypic mutational status of KLF1 mutation with the level of Hb F and Hb A2 in the patients of beta thalassemia and with the clinical data (frequency of blood transfusions).

CONTACTS AND LOCATIONS:
Overall Officials: Reem Abd Elkhalek Mohamed, lecturer, Study Director — Assiut University; Hebatallah Ahmed, lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Siatecka M, Bieker JJ. The multifunctional role of EKLF/KLF1 during erythropoiesis. Blood. 2011 Aug 25;118(8):2044-54. doi: 10.1182/blood-2011-03-331371. Epub 2011 May 25. PMID 21613252
- [Background] Tallack MR, Perkins AC. Three fingers on the switch: Kruppel-like factor 1 regulation of gamma-globin to beta-globin gene switching. Curr Opin Hematol. 2013 May;20(3):193-200. doi: 10.1097/MOH.0b013e32835f59ba. PMID 23474875
- [Background] Elagooz R, Dhara AR, Gott RM, Adams SE, White RA, Ghosh A, Ganguly S, Man Y, Owusu-Ansah A, Mian OY, Gurkan UA, Komar AA, Ramamoorthy M, Gnanapragasam MN. PUM1 mediates the posttranscriptional regulation of human fetal hemoglobin. Blood Adv. 2022 Dec 13;6(23):6016-6022. doi: 10.1182/bloodadvances.2021006730. PMID 35667093
- [Background] Borg J, Papadopoulos P, Georgitsi M, Gutierrez L, Grech G, Fanis P, Phylactides M, Verkerk AJ, van der Spek PJ, Scerri CA, Cassar W, Galdies R, van Ijcken W, Ozgur Z, Gillemans N, Hou J, Bugeja M, Grosveld FG, von Lindern M, Felice AE, Patrinos GP, Philipsen S. Haploinsufficiency for the erythroid transcription factor KLF1 causes hereditary persistence of fetal hemoglobin. Nat Genet. 2010 Sep;42(9):801-5. doi: 10.1038/ng.630. Epub 2010 Aug 1. PMID 20676099
- [Background] Srivorakun H, Thawinan W, Fucharoen G, Sanchaisuriya K, Fucharoen S. Thalassemia and erythroid transcription factor KLF1 mutations associated with borderline hemoglobin A2 in the Thai population. Arch Med Sci. 2020 Aug 11;18(1):112-120. doi: 10.5114/aoms.2020.93392. eCollection 2022. PMID 35154532
- [Background] Waye JS, Eng B. Kruppel-like factor 1: hematologic phenotypes associated with KLF1 gene mutations. Int J Lab Hematol. 2015 May;37 Suppl 1:78-84. doi: 10.1111/ijlh.12356. PMID 25976964
- [Background] Hariharan P, Colah R, Ghosh K, Nadkarni A. Differential role of Kruppel like factor 1 (KLF1) gene in red blood cell disorders. Genomics. 2019 Dec;111(6):1771-1776. doi: 10.1016/j.ygeno.2018.11.032. Epub 2018 Dec 5. PMID 30529538
- [Background] Xie XM, Liu YN, Li J, Jiang F, Li DZ. A Kruppel-Like Factor 1 Gene Mutation Ameliorates the Severity of beta-Thalassemia: A Case Report. Hemoglobin. 2019 Mar;43(2):137-139. doi: 10.1080/03630269.2019.1607373. Epub 2019 May 21. PMID 31111750
- [Background] El-Beshlawy A, Youssry I. Prevention of hemoglobinopathies in Egypt. Hemoglobin. 2009;33 Suppl 1:S14-20. doi: 10.3109/03630260903346395. PMID 20001619
- [Result] Origa R. beta-Thalassemia. Genet Med. 2017 Jun;19(6):609-619. doi: 10.1038/gim.2016.173. Epub 2016 Nov 3. PMID 27811859